CLINICAL TRIAL: NCT05381740
Title: A Novel Brain Stimulation for Bimanual Motor Function and Control in Chronic Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ela B. Plow, Assistant Professor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-074
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: stroke; brain stimulation; TMS; Upper Limb; rehabilitation; MRI; CVA; neuromodulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: In a prospective randomized controlled trial, an anticipated 18 stroke survivors with chronic (≥6 months) upper limb impairment will receive real or sham stimulation to the non-stroke hemisphere (cHMC). Stimulation will be delivered in conjunction with upper limb rehabilitation for 2 days a week for 6 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be told they will receive brain stimulation, but will be given no indication as to whether they will receive real or sham stimulation. Investigators analyzing functional outcome data, neurophysiology data and MRI data will receive coded data that conceals the identity of the subject. Therapists involved in training patients will not know which type of rTMS the participant receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- cHMC rTMS + Upper Limb Training Training (Experimental): Real Repetitive Transcranial Magnetic Stimulation given to facilitate the Contralesional Higher Motor Cortices+ Upper Limb Training
  Interventions: Device: Novel rTMS Approach
- Sham rTMS + Upper Limb Training Training (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation over Contralesional Higher Motor Cortices+ Upper Limb Training
  Interventions: Device: Sham rTMS Approach

INTERVENTIONS:
Device: Novel rTMS Approach — Participants in this arm will receive rTMS-based facilitation of the contralesional higher motor cortices located in the non-stroke hemisphere before the start of each rehabilitation session. High-frequency rTMS (5Hz) will be delivered using 42 10 second trains of 50 pulses each (total 2100 pulses) for a period of 22 minutes. Immediately after the completion of rTMS, participants will undergo therapist-guided upper limb therapy for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks for a total of 12 sessions.
  Arms: cHMC rTMS + Upper Limb Training Training
Device: Sham rTMS Approach — Participants in this arm will receive sham rTMS given over the contralesional higher motor cortices located in the non-stroke hemisphere before the start of each rehabilitation session. Immediately after the completion of sham rTMS, participants will undergo therapist-guided upper limb therapy for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks for a total of 12 sessions.
  Arms: Sham rTMS + Upper Limb Training Training

SUMMARY:
The long-term goal of this project is to develop and test upper Iimb rehabilitation interventions that can improve bimanual motor function, or the ability to use both arms and hands together, for stroke survivors with moderate to severe impairment.

This study will utilize a novel method of non-invasive brain stimulation in conjunction with upper limb training given for 12 visits over a period of 6 weeks.

The study will include the following site visits:

* Eligibility Screening and Informed Consent Visit
* Baseline testing (4 visits total): 1 visit each for MRI, upper limb and bimanual motor function test, bimanual motor control, and neurophysiology related to control of the upper limbs
* Repeat baseline testing (4 visits total) of MRI, upper limb and bimanual motor function test, bimanual motor control, and neurophysiology related to control of the upper limbs
* 12 intervention visits during which patients will receive upper limb therapy in conjunction with non-invasive brain stimulation
* Repeat testing (4 visits total) of MRI, upper limb and bimanual motor function test, bimanual motor control, and neurophysiology related to control of the upper limbs
* A follow-up visit 1 month after the completion of interventions

DETAILED DESCRIPTION:
In a pilot randomized controlled clinical trial, 18 stroke survivors more than 6 months after stroke onset, and have upper limb impairment will be enrolled. Participants will be randomized to receive a form of non-invasive brain stimulation called repetitive transcranial magnetic stimulation or rTMS or sham rTMS. Real or sham rTMS will be delivered over an area in the brain called the higher motor cortices within the stroke-unaffected hemisphere, cHMC for short. This area (cHMC) is important for using both arms and hands together, or bimanual motor function. Real or sham cHMC rTMS will be given prior to upper limb therapy twice a week for 6 weeks in the lab. The investigators will measure bimanual motor function and control twice at the beginning, once after the 6-week treatment and once at 1-month after treatment. The investigators will also test possible mechanisms related to the treatment using brain functional MRI and TMS twice at the beginning and once after 6-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 yrs
* ≥6 months since first clinical stroke
* Impairment of the paretic hand, indicated by a score of <= 11 out of 14 on the hand section of UEFM
* Sufficient range of motion in the wrist and fingers for functional task practice: have at least 10 degrees active wrist extension, 10 degrees active thumb abduction/extension, and 10 degrees active extension in at least 2 additional digits
* Sufficient active shoulder and elbow movement to volitionally position the paretic hand in the workspace for table-top task practice

Exclusion Criteria:

* Brainstem or cerebellar stroke
* Bilateral strokes or multiple strokes affecting sensorimotor structures
* Cognitive impairment (Mini-Mental State Examination <24)
* Severe impairment of the paretic hand that limits functional task practice (UEFM hand score < 4 out of 14)
* Severe spasticity (Modified Ashworth Scale >3) or upper limb contracture
* Occupational therapy or upper limb Botox completed ≤ 2 months prior
* Contraindications to TMS or MRI (e.g. metal implant in head, seizure history, cardiac pacemaker)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Bimanual Assessment Measure (BAM) | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks) and after end of 1 month of follow-up.
  Measure of the functional ability to perform 11 bimanual tasks scoring the spontaneous role of the affected hand, timing, and quality of movement.

SECONDARY OUTCOMES:
Change in Bimanual Grip Force Modulation Task | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks) and after end of 1 month of follow-up.
  Measure the ability to produce and maintain differing levels of force using hand dynamometers. This measurement represents patient's ability to perform independent tasks with each hand.
Change in ABILHAND | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks) and after end of 1 month of follow-up.
  ABILHAND assesses the participant's perception of bimanual ability by rating the difficulty of performing 23 bimanual activities without assistance on a 3 point ordinal scale (impossible, difficult, easy) This test has excellent reliability (ICC = 0.85-0.91).
Change in Upper Extremity Fugyl-Meyer Score (UEFM) | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks) and after end of 1 month of follow-up.
  Impairment will be measured using UEFM, one of the most widely used assessments in stroke. UEFM will serve as our primary outcome because it is sensitive to discerning the effects of rTMS/rehabilitation, and has excellent reliability (ICC= 0.97), consistency (Cronbach's α= 0.84) and validity. UEFM has a score ranging from 0-66 (0 meaning there is no movement of the paretic arm, and 66 meaning there is no functional limitation of the paretic arm.)
Change in Wolf Motor Function Test (WMFT) | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks) and after end of 1 month of follow-up.
  Functional ability to use the paretic upper limb in a variety of tasks will be assessed using WMFT. Time to complete each task will be noted and converted to rate (60/Performance Time (sec)), optimized for measurement in moderately/severely-impaired patients. Grip strength will also be recorded with WMFT.
Change Resting State Functional Magnetic Resonance Imaging(rsfMRI) | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks)
  Functional connectivity will assess the connectivity between cHMC and iM1 using temporal correlation of blood oxygneation level-dependent (BOLD) signal given as z-scores.
Change in excitability of cortical and corticospinal physiology (TMS) | Baseline (0 weeks and 2 weeks), after intervention(up to 7 weeks)
  Transcranial magnetic stimulation will be used to test crossed and uncrossed output from both hemispheres and will be measured as motor evoked potentials(MEPS) of the Extensor Digitorum Communis (EDC).

CONTACTS AND LOCATIONS:
Overall Officials: Ela Plow, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Lerner Research Institute, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haaland KY, Mutha PK, Rinehart JK, Daniels M, Cushnyr B, Adair JC. Relationship between arm usage and instrumental activities of daily living after unilateral stroke. Arch Phys Med Rehabil. 2012 Nov;93(11):1957-62. doi: 10.1016/j.apmr.2012.05.011. Epub 2012 May 24. PMID 22634230
- [Background] Sankarasubramanian V, Machado AG, Conforto AB, Potter-Baker KA, Cunningham DA, Varnerin NM, Wang X, Sakaie K, Plow EB. Inhibition versus facilitation of contralesional motor cortices in stroke: Deriving a model to tailor brain stimulation. Clin Neurophysiol. 2017 Jun;128(6):892-902. doi: 10.1016/j.clinph.2017.03.030. Epub 2017 Mar 21. PMID 28402865
- [Background] Liao WW, Whitall J, Wittenberg GF, Barton JE, McCombe Waller S. Not all brain regions are created equal for improving bimanual coordination in individuals with chronic stroke. Clin Neurophysiol. 2019 Aug;130(8):1218-1230. doi: 10.1016/j.clinph.2019.04.711. Epub 2019 May 13. PMID 31163366